CLINICAL TRIAL: NCT04087330
Title: Effects of Whole-body Vibration on Spasticity, Balance and Mobility in Spastic Hemiplegic Cerebral Palsy
Brief Title: Whole-body Vibration in Spastic Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00555 kainat Ameer
Record Dates: First submitted 2019-09-04; First posted 2019-09-12 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Cerebral Palsy; Spastic; Whole body vibration
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Experimental group (Experimental): Stretching, facilitation exercises with whole body vibration
  Interventions: Other: Group 1 Experimental group
- Group 2 Control group (Active Comparator): Stretching and facilitation exercises
  Interventions: Other: Group 2 Control group

INTERVENTIONS:
Other: Group 1 Experimental group — Stretching exercises for Achilles tendon, hamstrings, hip flexors and adductors of lower limbs, upper abdominal and pectoralis muscles.
  Facilitation of postural reactions, including: facilitation of righting, equilibrium and protective reactions from sitting on ball.
  Facilitation of standing and weight shift. Facilitation of standing balance by tilting the child from standing to different directions (forward, back-ward and side-way) using a balance board.
  Gait training: by forward, backward, and side-way walking between parallel bars.
  Whole body vibration.
  Arms: Group 1 Experimental group
Other: Group 2 Control group — Stretching exercises for Achilles tendon, hamstrings, hip flexors and adductors of lower limbs, upper abdominal and pectoralis muscles.
  Facilitation of postural reactions, including: facilitation of righting, equilibrium and protective reactions from sitting on ball.
  Facilitation of standing and weight shift. Facilitation of standing balance by tilting the child from standing to different directions (forward, back-ward and side-way) using a balance board.
  Gait training: by forward, backward, and side-way walking between parallel bars.
  Arms: Group 2 Control group

SUMMARY:
To target spasticity, balance and mobility whole body vibration exercises along with selected physical therapy is given to experimental group. Control group will receive only selected physical therapy that includes sstretching exercises, gait training, ffacilitation of postural reactions, ffacilitation of standing and weight shift and facilitation of standing balance by using a balance board.

DETAILED DESCRIPTION:
Cerebral palsy is the most common childhood disabilities affecting individual's posture and movement. Cerebral palsy is a disorder that causes activity limitations attributed to non-progressive disturbances of the foetal or infant brain that may also affect sensation, perception, cognition, communication, and behavior. Cerebral palsy (CP) results from damage to the developing central nervous system while in utero, during delivery, or during the first two years of life.

The most common movement disorder in Cerebral palsy is a spastic paresis, defined as a posture and movement-dependent tone regulation disorder.The most common signs of the disorder are spasticity, rigidity, muscle weakness, ataxia, balance and movement disorders. Compared to the typically developed children, these children have impaired sensation and increased muscle tone therefore they have trouble voluntarily controlling their muscles. Cerebral Palsy can be grouped based on the motor effects it has on the individual, these can include spastic Cerebral palsy or non-spastic Cerebral palsy. Spastic Cerebral Palsy is the most common type and is associated with tight or contracted muscles.

Cerebral Palsy is more prevalent in more deprived socio-economic populations. Cerebral palsy is a disease that globally has a prevalence of 2 to 3 cases per 1,000 live born neonates. An increase in the prevalence of CP was also seen in low birth weight survivors from the Mersey region of the United Kingdom for the same period. Pilot studies of severe mental retardation conducted in selected populations in Pakistan and India have reported extraordinarily high prevalence estimates in the range of 12-24 /1,000 Spasticity may be defined as a motor disorder characterised by a velocity-dependent exaggeration of stretch reflexes resulting from abnormal intraspinal processing of primary afferent input. The impaired sensation and increase in tone leads to wide range in movement dysfunction. About seventy to eighty percent of children with Cerebral Palsy demonstrate spastic clinical features. Many children with cerebral palsy (CP) have poor walking abilities and manipulation skills. One contributing factor to their problems with gait and reaching movement is poor balance control. Balance control is important as it helps a child to recover from unexpected balance disturbances.Currently, there are many options for the management of spasticity, balance disturbances and risk of fall that includes physical modalities, oral pharmacologic agents, peripheral injectables, intrathecal agents, and surgical interventions, however mostly physical therapy is commonly preferable treatment that includes stretching, NDT, Proprioceptive neuromuscular facilitations,strength training and gait training.

Dynamic mechanical loading of the skeleton is an arduous task and troublesome to induce in children who suffer from severe cerebral palsy. The lack of dynamic weight bearing in this population predisposes them to reduced bone mineral density (BMD) and pre-mature osteoporosis. These children are also more prone to muscle weakness, which contributes to pain, deformity and functional loss. Whole-body vibration training was proposed as a new therapeutic modality for the treatment of the gross motor function, balance and functional performance Whole body vibration (WBV), for which the participant stands on a vibrating platform, delivers low-frequency, low-amplitude mechanical stimuli that enter the human body via the feet. The vibrations stimulate the muscle spindles and alpha motor neuron sending nerve impulses to initiate muscle contractions according to the tonic vibration reflex. Compared to the repetitive passive movement, this WBV protocol adds a muscle strengthening component to the anti-spastic effects. Activity restrictions in spastic cerebral palsy are mainly due to poor postural control. Many interventions like resisting exercises, therapeutic horseback riding, electrical stimulations leads to short term posture and balance improvement. Training using vibration platforms adjunct to exercise has shown to be effective in increasing strength resulting in improved balance and coordination. Whole body vibration has shown to be effective in reducing lower limb spasticity after first application of WBV with a vibration frequency of 12 Hz to 18 Hz ( 2-3 m of amplitude ) for 9 minutes and a significant decrease in tone is observed and even the functional mobility and balance is improved.. During all of the vibration-training sessions, the children will wear the gymnastic shoes to standardize the damping of the vibration due to footwear.

There is paucity in the literature regarding evidence for the safe and effective use of vibration intervention in children with or without pathology and has great effects in spasticity, mobility and improving balance.Chia-Ling Chen concluded that the WBV is an effective intervention for controlling spasticity and improving ambulation. Villarreal et al.showed that 20-week WBV therapy had positive effects on the balance of DS adolescents, although only under specific conditions, with vision and somatosensory input altered.

In previous studies high dosage of whole body vibration has both positive and negative effects. Because this type of treatment seems to improve bone health, The purpose of this intervention is to ensure functional independence in cerebral palsy patients. Whole Body Vibration Therapy has proven to be effective in improving balance by reducing spasticity and improving muscle strength. It is essential to explore new interventions for patients specially for cerebral palsy in whom functional independence is impaired thus their mobility is restricted leading to secondary complications. In my study my goal is to use combination of conventional physical therapy with whole body vibration which can control spasticity and enhance ambulatory performance.

ELIGIBILITY:
Inclusion Criteria:

* Ashworth scale score +1-3
* age between 6 and 13 years,
* able to accept and follow verbal instructions,
* Gross Motor Function Classification System [GMFCS] levels I-III),

Exclusion Criteria:

* unstable seizures, any treatment for spasticity or surgical procedures from 3 months (for botulinum toxin type A injections)
* Suffering from any other condition that interfered with physical activity.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth | Change from Baseline spasticity to 3 months
  It is used to check spasticity and consists of 6 grades from 0-4
6-Minute walking test (6MWT) | Change from Baseline mobility level to 3 months
  It is used to test mobility of participant. The 6-minute walk test (6MWT) is a standardized, self-paced walking test commonly used to assess functional ability in different populations.
Paediatric Balance Scale | Change from Baseline balance to 3 months
  The Pediatric Balance Scale (PBS), a modification of the BBS, was developed as a balance measure for children with mild to moderate motor impairments and has good test-retest and interrater reliability. The PBS is a 14-item, criterion-referenced measure and examines functional balance in the context of everyday tasks

SECONDARY OUTCOMES:
Timed Up and Go test (TUG) | Change from Baseline mobility and balance to 3 months
  TUG is a test used to assess a person's mobility. TUG measured the time required for an individual to stand up from a chair with armrests, walk 3 m, turn, walk back to the chair, and sit down.
Sit-To-Stand (STS) test | Change from Baseline mobility and balance to 3 months
  Sit to stand test is a reliable tool for measuring lower limb functional strength and balance ability.

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Ghous, MSNMPT*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng HY, Ju YY, Chen CL, Chuang LL, Cheng CH. Effects of whole body vibration on spasticity and lower extremity function in children with cerebral palsy. Hum Mov Sci. 2015 Feb;39:65-72. doi: 10.1016/j.humov.2014.11.003. Epub 2014 Nov 24. PMID 25461434
- [Background] Dickin DC, Faust KA, Wang H, Frame J. The acute effects of whole-body vibration on gait parameters in adults with cerebral palsy. J Musculoskelet Neuronal Interact. 2013 Mar;13(1):19-26. PMID 23445911
- [Background] Saquetto M, Carvalho V, Silva C, Conceicao C, Gomes-Neto M. The effects of whole body vibration on mobility and balance in children with cerebral palsy: a systematic review with meta-analysis. J Musculoskelet Neuronal Interact. 2015 Jun;15(2):137-44. PMID 26032205
- [Background] Unger M, Jelsma J, Stark C. Effect of a trunk-targeted intervention using vibration on posture and gait in children with spastic type cerebral palsy: a randomized control trial. Dev Neurorehabil. 2013;16(2):79-88. doi: 10.3109/17518423.2012.715313. PMID 23477461
- [Background] Matute-Llorente A, Gonzalez-Aguero A, Gomez-Cabello A, Vicente-Rodriguez G, Casajus Mallen JA. Effect of whole-body vibration therapy on health-related physical fitness in children and adolescents with disabilities: a systematic review. J Adolesc Health. 2014 Apr;54(4):385-96. doi: 10.1016/j.jadohealth.2013.11.001. Epub 2014 Jan 1. PMID 24388109
- [Background] Yeargin-Allsopp M, Van Naarden Braun K, Doernberg NS, Benedict RE, Kirby RS, Durkin MS. Prevalence of cerebral palsy in 8-year-old children in three areas of the United States in 2002: a multisite collaboration. Pediatrics. 2008 Mar;121(3):547-54. doi: 10.1542/peds.2007-1270. PMID 18310204